CLINICAL TRIAL: NCT00041938
Title: Warfarin Versus Aspirin in Reduced Cardiac Ejection Fraction (WARCEF) Trial
Acronym: WARCEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Shunichi Homma, Margaret Milliken Hatch Professor of Medicine at the New York-Presbyterian Hospital at the Columbia University Medical Center (In Biomedical Engineering), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAC1093; U01NS039143-01 (NIH); R01NS39154; CRC
Record Dates: First submitted 2002-07-19; First posted 2002-07-22 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Heart Disease; Stroke; Ischemic Heart Disease; Myocardial Infarction
Keywords: heart disease; stroke; ischemic heart disease; myocardial infarction; atrial fibrillation; low ejection fraction; cardiac failure; aspirin; Warfarin; anticoagulant
MeSH Terms: conditions — Heart Diseases; Stroke; Myocardial Ischemia; Myocardial Infarction; Atrial Fibrillation; Heart Failure | interventions — Aspirin; Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin (Active Comparator): Aspirin: 325 mg per day
  Interventions: Drug: aspirin
- warfarin (Active Comparator): Warfarin: International Normalized Ratio (INR) 2.5-3.0; target INR 2.75
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: aspirin — 325 mg per day
  Arms: aspirin
Drug: Warfarin — INR 2.5-3.0; target INR 2.75
  Arms: warfarin

SUMMARY:
The purpose of this study is to determine which of two treatments, Warfarin or aspirin, is better for preventing death and stroke in patients with poor heart function.

We are now transitioning into the sub-analysis part of the WARCEF patient data.

The study has recently completed data analysis for its Primary Aim. All randomized patients have completed their follow up. All study related procedure as per the protocol has been completed. We are now in the extension phase of the study to obtain more patient data to address further aims of the study. No new procedures are performed and data already in place at the sites will be collected (EKG and echocardiograms).

The aims for this study extension are:

* To assess progression of cardiac dysfunction over time among heart failure patients
* To correlate prognosis with cardiac dysfunction

DETAILED DESCRIPTION:
Warfarin has proven effective in patients with ischemic heart disease, especially in the reduction of stroke, death and re-infarction following myocardial infarction, and in the reduction of stroke in atrial fibrillation. Warfarin is the most promising unstudied intervention in patients with cardiac failure. This randomized, double-blind, multi-center study will define optimal antithrombotic therapy for patients with cardiac (heart) failure and patients with low ejection fraction (EF). EF is the proportion of left ventricular volume emptied during systole. It reliably measures left ventricular systolic function.

With the rapidly increasing numbers of elderly patients with heart failure, this study has important public health implications. The study will determine which of two commonly used treatments Warfarin, an anticoagulant, or aspirin, a drug which affects platelet function is better for preventing death and stroke in patients with low ejection fraction.

ELIGIBILITY:
Inclusion Criteria

* Cardiac EF <=35% by radionuclide ventriculography, left ventriculography or quantitive echocardiographic measurement or an echocardiographic Wall Motion Index of <=1.2, within three months of enrollment. The patient's clinical cardiac state at enrollment should be similar to their state at the time of the qualifying echocardiogram. The qualifying left ventricular function measurement must be obtained at least three months after an MI, coronary bypass grafting, PTCA, and at least one month after pacemaker insertion. Patients scheduled for mitral valve repair should have qualifying echo after surgery.
* Modified Rankin score <=4.
* Patient must be taking ACE inhibitors. If intolerant of ACE inhibitor, patient must be on angiotensin II receptor blockers or hydralazine and nitrates.
* Patient is able to follow an outpatient protocol (requiring monthly blood tests and clinic visits every four months for the duration of the study) and is available by telephone.
* Patient understands the purpose and requirements of the study, can make him/herself understood, and has provided informed consent.
* Patients with recent stroke or TIA within twelve (12) months will be eligible to be included in the recent stroke (RS) subgroup.
* Chronic CHF patients (NYHA I * IV) admitted to the hospital can be randomized prior to discharge if the patient is stable, taking oral medications for 24 hours and ambulatory at the time of discharge. Stable New York Heart Association Class IV patients will be eligible for randomization.

Exclusion Criteria

* The presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal AF, mechanical valve, endocarditis, intracardiac mobile or pedunculated thrombus, and valvular vegetation.
* Cyanotic congenital heart disease, Eisenmenger's syndrome.
* Decompensated heart failure.
* Cardiac surgery, angioplasty, or MI within the past 3 months prior to randomization.
* A contraindication to the use of either warfarin or aspirin, e.g. active peptic ulcer disease, active bleeding diathesis, platelets <100,000*, hematocrit <30, INR >1.3 (if not on warfarin), clotting factor abnormality that increases the risk of bleeding, alcohol or substance abuse, severe gait instability, cerebral hemorrhage, systemic hemorrhage within the past year, severe liver impairment (AST >3x normal*, cirrhosis), any condition requiring regular use of non-steroidal anti-inflammatory agents, allergy to aspirin or warfarin, uncontrolled severe hypertension (systolic pressure >180 mm Hg or diastolic pressure > 110 mm Hg), positive stool guaiac not attributable to hemorrhoids, creatinine >3.0*. *on most recent test done within 30 days prior to randomization
* Patient needs continuing therapy with intravenous heparin or low molecular weight heparin or a specific antiplatelet agent.
* Dementia or psychiatric or physical problem that prevents the patient from following an outpatient program reliably.
* Comorbid conditions that may limit survival to less than five years.
* Pregnancy, or female of childbearing potential who is not sterilized or is not using a medically accepted form of contraception* (see procedure manual). *A pregnancy test is required for all women of childbearing age.
* Enrollment in another study that would conflict with WARCEF.
* Hospitalization for new diagnosis of onset CHF within the past one month or carotid endarterectomy or pacemaker insertion within the past one month prior to randomization .
* Person under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2305 (Actual)
Dates: Start 2002-10; Primary Completion 2011-08 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shunichi Homma, M.D., Principal Investigator — Principal Cardiologist, Associate Chief, Division of Cardiology, and Director, Echocardiography Laboratories Professor of Medicine; Seamus Thompson, PhD, Principal Investigator — Statistical PI: Clinical Professor of Biostatistics and Neurology
Locations (64):
- United States (54):
  - Southern Arizona Veterans Affairs Medical Center, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Santa Clara Medical Center, Santa Clara, California
  - West Los Angeles Veterans Affairs Medical Center, West Los Angeles, California
  - Denver Health Medical Center, Denver, Colorado
  - Denver Veterans Affairs Medical Center, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Mayo Clinic Transplant Center, Jacksonville, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Jackson Memorial Hospital/U. of Miami, Miami, Florida
  - Mercy Research Institute, Miami, Florida
  - Cardiovascular Consultants of South Florida, Tamarac, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Methodist Heart, Lung and Vascular Institute, Peoria, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Louisville Veterans Affairs Medical Center, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Gulf Regional Research, LLC, Metairie, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Lahey Clinic, Burlington, Massachusetts
  - Veterans Affairs Medical Center, Detroit, Michigan
  - Mercy Health Partners, Muskegon, Michigan
  - Reno Veterans Affairs Medical Center, Reno, Nevada
  - Concord Hospital, Concord, New Hampshire
  - UMDNJ - New Brunswick, New Brunswick, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Albany Medical College, Albany, New York
  - Buffalo General Hospital, Buffalo, New York
  - Kaleida Health Millard Fillmore Hospital, Buffalo, New York
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University, New York Presbyterian Hospital PH 3-342, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Northport Veterans Affairs Medical Center, Northport, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Oklahoma City Veterans Affairs Medical Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Tri-State Medical Group Cardiology, Beaver, Pennsylvania
  - Sewickley Valley Medical Group, Cardiology, Leetsdale, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Black Hills Health Care System, Fort Meade, South Dakota
  - Brooke Army Medical Center MCHE - MDC Cardiology Service, Fort Sam Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center-MEDVAMC, Houston, Texas
  - Salem VAMC, Salem, Virginia
  - Huntington Veterans Affairs Medical Center, Huntington, West Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, Wisconsin
- Canada (10):
  - Center for Neurologic Research, Lethbridge, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Etobicoke Cardiac Research Centre, Rexdale, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Derived] Corica B, Romiti GF, Simoni AH, Mei DA, Bucci T, Thompson JLP, Qian M, Homma S, Proietti M, Lip GYH; WARCEF Investigators. Educational status affects prognosis of patients with heart failure with reduced ejection fraction: A post-hoc analysis from the WARCEF trial. Eur J Clin Invest. 2024 May;54(5):e14152. doi: 10.1111/eci.14152. Epub 2024 Jan 11. PMID 38205865
- [Derived] Lee TC, Qian M, Liu Y, Graham S, Mann DL, Nakanishi K, Teerlink JR, Lip GYH, Freudenberger RS, Sacco RL, Mohr JP, Labovitz AJ, Ponikowski P, Lok DJ, Matsumoto K, Estol C, Anker SD, Pullicino PM, Buchsbaum R, Levin B, Thompson JLP, Homma S, Di Tullio MR; WARCEF Investigators. Cognitive Decline Over Time in Patients With Systolic Heart Failure: Insights From WARCEF. JACC Heart Fail. 2019 Dec;7(12):1042-1053. doi: 10.1016/j.jchf.2019.09.003. PMID 31779926
- [Derived] Teerlink JR, Qian M, Bello NA, Freudenberger RS, Levin B, Di Tullio MR, Graham S, Mann DL, Sacco RL, Mohr JP, Lip GYH, Labovitz AJ, Lee SC, Ponikowski P, Lok DJ, Anker SD, Thompson JLP, Homma S; WARCEF Investigators. Aspirin Does Not Increase Heart Failure Events in Heart Failure Patients: From the WARCEF Trial. JACC Heart Fail. 2017 Aug;5(8):603-610. doi: 10.1016/j.jchf.2017.04.011. PMID 28774396
- [Derived] Di Tullio MR, Qian M, Thompson JL, Labovitz AJ, Mann DL, Sacco RL, Pullicino PM, Freudenberger RS, Teerlink JR, Graham S, Lip GY, Levin B, Mohr JP, Buchsbaum R, Estol CJ, Lok DJ, Ponikowski P, Anker SD, Homma S; WARCEF Investigators. Left Ventricular Ejection Fraction and Risk of Stroke and Cardiac Events in Heart Failure: Data From the Warfarin Versus Aspirin in Reduced Ejection Fraction Trial. Stroke. 2016 Aug;47(8):2031-7. doi: 10.1161/STROKEAHA.116.013679. Epub 2016 Jun 28. PMID 27354224
- [Derived] Freudenberger RS, Cheng B, Mann DL, Thompson JL, Sacco RL, Buchsbaum R, Sanford A, Pullicino PM, Levin B, Teerlink JR, Graham S, Mohr JP, Labovitz AJ, Di Tullio MR, Lip GY, Estol CJ, Lok DJ, Ponikowski P, Anker SD, Homma S; WARCEF Investigators. The first prognostic model for stroke and death in patients with systolic heart failure. J Cardiol. 2016 Aug;68(2):100-3. doi: 10.1016/j.jjcc.2015.09.014. Epub 2015 Nov 6. PMID 26549533
- [Derived] Homma S, Thompson JL, Qian M, Ye S, Di Tullio MR, Lip GY, Mann DL, Sacco RL, Levin B, Pullicino PM, Freudenberger RS, Teerlink JR, Graham S, Mohr JP, Labovitz AJ, Buchsbaum R, Estol CJ, Lok DJ, Ponikowski P, Anker SD; WARCEF Investigators. Quality of anticoagulation control in preventing adverse events in patients with heart failure in sinus rhythm: Warfarin versus Aspirin in Reduced Cardiac Ejection Fraction trial substudy. Circ Heart Fail. 2015 May;8(3):504-9. doi: 10.1161/CIRCHEARTFAILURE.114.001725. Epub 2015 Apr 7. PMID 25850425
- [Derived] Shaffer JA, Thompson JL, Cheng B, Ye S, Lip GY, Mann DL, Sacco RL, Pullicino PM, Freudenberger RS, Graham S, Mohr JP, Labovitz AJ, Estol CJ, Lok DJ, Ponikowski P, Anker SD, Di Tullio MR, Homma S; WARCEF Investigators. Association of quality of life with anticoagulant control in patients with heart failure: the Warfarin and Aspirin in Reduced Cardiac Ejection Fraction (WARCEF) trial. Int J Cardiol. 2014 Dec 15;177(2):715-7. doi: 10.1016/j.ijcard.2014.10.012. No abstract available. PMID 25456692
- [Derived] Homma S, Thompson JL, Sanford AR, Mann DL, Sacco RL, Levin B, Pullicino PM, Freudenberger RS, Teerlink JR, Graham S, Mohr JP, Massie BM, Labovitz AJ, Di Tullio MR, Gabriel AP, Lip GY, Estol CJ, Lok DJ, Ponikowski P, Anker SD; WARCEF Investigators. Benefit of warfarin compared with aspirin in patients with heart failure in sinus rhythm: a subgroup analysis of WARCEF, a randomized controlled trial. Circ Heart Fail. 2013 Sep 1;6(5):988-97. doi: 10.1161/CIRCHEARTFAILURE.113.000372. Epub 2013 Jul 23. PMID 23881846
- [Derived] Homma S, Thompson JL, Pullicino PM, Levin B, Freudenberger RS, Teerlink JR, Ammon SE, Graham S, Sacco RL, Mann DL, Mohr JP, Massie BM, Labovitz AJ, Anker SD, Lok DJ, Ponikowski P, Estol CJ, Lip GY, Di Tullio MR, Sanford AR, Mejia V, Gabriel AP, del Valle ML, Buchsbaum R; WARCEF Investigators. Warfarin and aspirin in patients with heart failure and sinus rhythm. N Engl J Med. 2012 May 17;366(20):1859-69. doi: 10.1056/NEJMoa1202299. Epub 2012 May 2. PMID 22551105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited 2305 patients at 176 sites in 11 countries, between 10/1/2002 and 1/31/2010.
Pre-assignment Details: Intent-to-treat trial - all randomized patients followed and analyzed.
Groups:
- Aspirin: Aspirin : 325 mg per day
- Warfarin: Warfarin : International Normalized Ratio (INR) 2.5-3.0; target INR 2.75
Period: Overall Study
Arm/Group | Aspirin | Warfarin
Started | 1163 | 1142
Completed Follow-up | 761 | 745
Primary Endpoint | 320 | 302
Only Vital Status Known | 44 | 46
Lost to Follow-up | 18 | 17
Withdrew Consent | 20 | 14
Completed | 1125 | 1111
Not Completed | 38 | 31

BASELINE CHARACTERISTICS:
Groups:
- Warfarin: Warfarin : INR 2.5-3.0; target INR 2.75
- Total: Total of all reporting groups
Arm/Group | Aspirin | Warfarin | Total
Number analyzed (Participants) | 1163 | 1142 | 2305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 732 | 706 | 1438
  >=65 years | 431 | 436 | 867
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11.1) | 61 (11.6) | 61 (11.3)
Sex/Gender, Customized [Number; unit: participants]
  Male | 936 | 904 | 1840
  Female | 224 | 236 | 460
  Unknown | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  North America | 546 | 573 | 1119
  Europe | 567 | 527 | 1094
  Argentina | 50 | 42 | 92

OUTCOME MEASURES:

1. Primary Outcome: Event Rate Per 100 Patient Years for Composite Endpoint of Ischemic Stroke, Intracerebral Hemorrhage, or Death
Description: The time, in years, from randomization to the first to occur of ischemic stroke, intracerebral hemorrhage, or death, up to a maximum of 6 years. Event rate per 100 patient years = 100*(number of subjects with event)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization until the date of the first to occur of ischemic stroke, intracerebral hemorrhage, or death, up to 6 years
Population: Intent-to-treat analysis: all enrolled patients were analyzed.
Measure: Number; unit: events per 100 patient-years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient-years | 7.93 | 7.47
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; The primary null hypothesis: time to first event in the composite primary endpoint does not differ significantly between warfarin and aspirin. The original target sample size was 2860, providing 89% power for a log-rank test with two-sided alpha .05, assuming a hazard rate reduction of 17.82% in either group compared with the other, after adjustment for use of beta-blockers and allowance for discontinuation of therapy, dropout, and crossover. The final sample of 2305 patients yielded 69% power; Test type: Superiority or Other; p = 0.40, Regression, Cox — The primary null hypotheses was tested at two-tailed alpha=0.05. A Haybittle-Peto interim monitoring procedure was performed with stopping boundaries for the interim analyses corresponding to a nominal two-tailed P value of 0.001; Cox models stratified by site, New York Heart Association class (I vs. II-IV), and status w/ respect to recent stroke or Transient Ischemic Attack; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.79 to 1.10] — Hazard ratio is for comparison of warfarin vs. aspirin. Warfarin represents the numerator and aspirin represents the denominator of the hazard ratio

2. Secondary Outcome: Event Rate Per 100 Patient-years for Composite Endpoint of Hospitalization for Heart Failure, Myocardial Infarction, Ischemic Stroke, Intracerebral Hemorrhage, or Death.
Description: The time, in years, from date of randomization to the date of the first to occur of hospitalization for heart failure, myocardial infarction, ischemic stroke, intracerebral hemorrhage, or death, up to 6 years.
  Event rate per 100 patient years = 100*(number of subjects with event)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From randomization to the first to occur of hospitalization for heart failure, myocardial infarction, ischemic stroke, intracerebral hemorrhage, or death, up to a maximum of 6 years.
Population: Intent-to-treat analysis: all enrolled patients were analyzed.
Measure: Number; unit: events per 100 patient-years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient-years | 12.15 | 12.70
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Secondary null hypothesis: time to first event in the composite secondary endpoint does not differ significantly between warfarin and aspirin. This was tested at prespecified alpha = 0.05 level, two-tailed; Test type: Superiority or Other; p = 0.33, Regression, Cox — Secondary null hypothesis was tested at two-tailed alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.93 to 1.23] — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Event Rate Per 100 Patient-years for Ischemic Stroke
Description: Time, in years, from date of randomization to date of ischemic stroke component of primary composite outcome, up to 6 years. Event rate per 100 patient years = 100*(number of subjects with ischemic stroke)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization to date of ischemic stroke component of primary composite outcome, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: rate per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
rate per 100 patient years | 1.36 | 0.72
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Null hypothesis: there is no difference between warfarin and aspirin in time to ischemic stroke, adjusting for competing risks of death and intracerebral hemorrhage; Test type: Superiority or Other; p = 0.005, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.33 to 0.82] — [estimate comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Event Rate Per 100 Patient-years for Intracerebral Hemorrhage
Description: Time, in years, from date of randomization to date of intracerebral hemorrhage component of primary composite outcome. Event rate per 100 patient years = 100*(number of subjects with intracerebral hemorrhage)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization to date of intracerebral hemorrhage component of primary composite outcome, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: rate per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
rate per 100 patient years | 0.05 | 0.12
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Null hypothesis: there is no difference between warfarin and aspirin in time to intracerebral hemorrhage, adjusting for competing risks of death and ischemic stroke; Test type: Superiority or Other; p = 0.35, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 2.22, 95% CI [0.43 to 11.66]

5. Other Pre Specified Outcome: Event Rate Per 100 Patient-years for Death
Description: Time, in years, from date of randomization to date of death component of primary composite outcome. Event rate per 100 patient years = 100*(number of subjects who died)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization to date of death component of primary composite outcome, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: events per 100 patient-years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient-years | 6.52 | 6.63
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Test type: Superiority or Other; p = 0.91, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.85 to 1.20] — [estimate comment as in outcome 1, analysis 1]

6. Other Pre Specified Outcome: Event Rate Per 100 Patient Years of Myocardial Infarction Component of Secondary Composite Outcome
Description: Time, in years, from date of randomization to date of myocardial infarction, up to 6 years. Includes only myocardial infarctions that occurred during follow-up, before any heart failure hospitalization. Event rate per 100 patient years = 100*(number of subjects with myocardial infarction)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization to date of myocardial infarction component of secondary composite outcome, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: events per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient years | 0.87 | 0.80
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Null hypothesis: there is no difference between warfarin and aspirin in time to myocardial infarction, adjusting for competing risks of heart failure hospitalization, ischemic stroke, intracerebral hemorrhage, and death; Test type: Superiority or Other; p = 0.93, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.58 to 1.64] — [estimate comment as in outcome 1, analysis 1]

7. Other Pre Specified Outcome: Event Rate Per 100 Patient Years of Heart Failure Hospitalization Component of Secondary Composite Outcome.
Description: Time, in years, from date of randomization to date of heart failure hospitalization, up to 6 years. Includes hospitalizations for heart failure during follow-up that were not preceded by myocardial infarction. Event rate per 100 patient years = 100*(number of subjects with heart failure hospitalization)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization to date of heart failure hospitalization component of secondary composite outcome, up to 6 years
Population: Intent-to-treat.
Measure: Number; unit: events per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient years | 5.67 | 6.79
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Null hypothesis: there is no difference between warfarin and aspirin in time to heart failure hospitalization, adjusting for competing risks of myocardial infarction, ischemic stroke, intracerebral hemorrhage, and death; Test type: Superiority or Other; p = 0.053, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.998 to 1.47]

8. Other Pre Specified Outcome: Event Rate Per 100 Patient Years of Ischemic Stroke Component of Secondary Composite Outcome
Description: Ischemic stroke component of secondary composite endpoint. Includes only ischemic strokes that were not preceded by a myocardial infarction or heart failure hospitalization. The number of ischemic strokes that are components of the secondary outcome does not therefore match the number of ischemic strokes that are components of the primary outcome. Event rate per 100 patient years = 100*(number of subjects with ischemic stroke)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1)of all randomized patients / 365.25.
Time Frame: From date of randomization to date of ischemic stroke component of secondary composite outcome, up to 6 years
Population: Intent-to-treat.
Measure: Number; unit: events per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient years | 1.14 | 0.57
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Null hypothesis: there is no difference between warfarin and aspirin in time to ischemic stroke, adjusting for competing risks of myocardial infarction, heart failure hospitalization, death and intracerebral hemorrhage; Test type: Superiority or Other; p = 0.03, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.32 to 0.96]

9. Other Pre Specified Outcome: Event Rate Per 100 Patient Years of Intracerebral Hemorrhage Component of Secondary Composite Outcome
Description: Time, in years, from date of randomization to date of intracerebral hemorrhage component of secondary composite outcome. Includes only intracerebral hemorrhages not preceded by myocardial infarction or heart failure hospitalization. Event rate per 100 patient years = 100*(number of subjects with intracerebral hemorrhage)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization to date of intracerebral hemorrhage component of secondary composite outcome, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: events per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient years | 0.06 | 0.11
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Null hypothesis: there is no difference between warfarin and aspirin in time to intracerebral hemorrhage, adjusting for competing risks of myocardial infarction, heart failure hospitalization, ischemic stroke, and death; Test type: Superiority or Other; p = 0.51, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 1.77, 95% CI 2-sided [0.32 to 9.88] — [estimate comment as in outcome 1, analysis 1]

10. Other Pre Specified Outcome: Event Rate Per 100 Patient Years of Death Component of Secondary Composite Outcome
Description: Time, in years, from randomization to death component of secondary composite outcome. This measure counts only deaths that were not preceded by heart failure hospitalization, myocardial infarction, ischemic stroke, or intracerebral hemorrhage. Event rate per 100 patient years = 100*(number of subjects who died)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization to date of death component of secondary composite outcome, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: events per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient years | 4.41 | 4.43
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Test type: Superiority or Other; p = 0.83, Regression, Cox; Cause-specific Cox model, stratified by site, NYHA class (I vs. II, III, or IV), and prior stroke or TIA status; Hazard Ratio (HR) = 1.03, 95% CI [0.81 to 1.30]

11. Other Pre Specified Outcome: Rate Per 100 Patient Years of Major Hemorrhage
Description: Rate/100 patient-years of major hemorrhage. Includes all major hemorrhages in any patient. Major hemorrhage was defined as intracerebral, epidural, subdural, subarachnoid, spinal intramedullary, or retinal hemorrhage; any other bleeding causing a decline in the hemoglobin level of more than 2 g per deciliter in 48 hours; or bleeding requiring transfusion of 2 or more units of whole blood, hospitalization, or surgical intervention. Event rate per 100 patient years = 100*(number of major hemorrhage events)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1) of all randomized patients / 365.25.
Time Frame: From date of randomization until end of scheduled follow-up, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: events per 100 patient years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient years | 0.87 | 1.78
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Test type: Superiority or Other; p < 0.001, Regression, Poisson; Rate ratio = 2.05, 95% CI 2-sided [1.36 to 3.12] — The warfarin arm represents the numerator and the aspirin arm represents the denominator of the rate ratio

12. Other Pre Specified Outcome: Rate Per 100 Patient-years of Minor Hemorrhage.
Description: Rate per 100 patient years of minor hemorrhage. Includes all minor hemorrhages. Minor hemorrhage was defined as any non-major hemorrhage. Event rate per 100 patient years = 100*(number of minor hemorrhage events)/patient-years of follow-up. Patient years of follow-up = sum(date of conclusion of follow-up - date of randomization + 1)of all randomized patients / 365.25.
Time Frame: From date of randomization until the end of scheduled follow-up, up to 6 years
Population: Intent-to-treat
Measure: Number; unit: events per 100 patient-years
Arm/Group | Aspirin | Warfarin
Number analyzed (Participants) | 1163 | 1142
events per 100 patient-years | 7.34 | 11.6
Statistical Analysis 1: Comparison: Aspirin vs Warfarin; Test type: Superiority or Other; p < 0.001, Regression, Poisson; Rate ratio = 1.56, 95% CI [1.34 to 1.81] — Warfarin group represents the numerator and aspirin group represents denominator of rate ratio

ADVERSE EVENTS:
Arm/Group | Aspirin | Warfarin
Serious Adverse Events (participants affected / at risk) | 617/1163 | 632/1142
Other Adverse Events (participants affected / at risk) | 749/1163 | 799/1142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=1163) | Warfarin (N=1142)
ALLERGY/IMMUNOLOGY: Other (General disorders) | 1 (1) | 1 (1)
Laryngeal edema/Allergic reaction/Anaphylaxis/Angioedema/Rash (General disorders) | 4 (4) | 2 (2)
Blood dyscrasia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
BLOOD/BONE MARROW: Other (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Thrombocytopenia/Anemia/Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 12 (12)
Atrial fibrillation/Atrial flutter/Supraventricular tachycardia (Cardiac disorders) | 56 (67) | 35 (45)
Bradycardia (Cardiac disorders) | 6 (6) | 6 (6)
CARDIAC ARRHYTHMIA: Other (Cardiac disorders) | 7 (7) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 7 (8) | 15 (17)
Ventricular tachycardia (Cardiac disorders) | 24 (33) | 39 (46)
Acute cardiac failure/CHF/Pulmonary edema (Cardiac disorders) | 209 (432) | 243 (506)
AICD firing/discharge (Cardiac disorders) | 16 (21) | 20 (21)
Angina/Chest pain (Cardiac disorders) | 70 (105) | 88 (148)
CARDIAC GENERAL: Other (Cardiac disorders) | 16 (18) | 16 (19)
Malignant hypertension (Cardiac disorders) | 3 (3) | 7 (7)
Myocardial infarction/Acute Coronary Syndrome (Cardiac disorders) | 48 (60) | 50 (59)
Pulmonary embolism (Cardiac disorders) | 6 (6) | 5 (5)
CONSTITUTIONAL SYMPTOMS: Other (General disorders) | 7 (7) | 1 (1)
DERMATOLOGY/SKIN: Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Grade 4 dermatologic manifestations (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Diabetes mellitus and its complications (Endocrine disorders) | 26 (35) | 22 (35)
ENDOCRINE: Other (Endocrine disorders) | 2 (2) | 1 (1)
Gastrointestinal disturbance/Diarrhea/Jaundice/Nausea/Stomach pain/Etc. (Gastrointestinal disorders) | 54 (70) | 66 (82)
GASTROINTESTINAL: Other (Gastrointestinal disorders) | 25 (31) | 17 (18)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 3 (3) | 3 (3)
HEPATOBILIARY/PANCREAS: Other (Hepatobiliary disorders) | 3 (3) | 5 (7)
Infection/Sepsis/Fever (Infections and infestations) | 66 (79) | 79 (97)
LYMPHATICS: Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Peripheral edema (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
MALIGNANCY: Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (24) | 20 (24)
Metabolic disturbance/Gout (Metabolism and nutrition disorders) | 14 (15) | 16 (17)
METABOLIC/LABORATORY: Other (Metabolism and nutrition disorders) | 12 (14) | 10 (11)
MUSCULOSKELETAL/SOFT TISSUE: Other (Musculoskeletal and connective tissue disorders) | 39 (43) | 29 (32)
Visceral necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Convulsions/Seizures (Nervous system disorders) | 6 (6) | 5 (10)
NEUROLOGY: Other (Nervous system disorders) | 8 (8) | 7 (7)
Stroke or TIA (Nervous system disorders) | 13 (16) | 15 (16)
Syncope/Pre-syncope (Nervous system disorders) | 41 (48) | 68 (83)
OCULAR/VISUAL: Other (Eye disorders) | 5 (7) | 3 (5)
Drug abuse (General disorders) | 3 (3) | 1 (1)
OTHER: Other (General disorders) | 19 (23) | 32 (33)
Pregnancy (General disorders) | 0 (0) | 1 (1)
Suicide attempt/Psychiatric disorder (General disorders) | 16 (16) | 10 (10)
PAIN: Other (General disorders) | 14 (15) | 13 (20)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (9)
Pulmonary disease/Pneumonia/Bronchitis/Asthma/Breathing difficulties (Respiratory, thoracic and mediastinal disorders) | 87 (133) | 79 (100)
PULMONARY/UPPER RESPIRATORY: Other (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Acute renal failure/Proteinuria (Renal and urinary disorders) | 28 (32) | 33 (36)
RENAL/GENITOURINARY: Other (Renal and urinary disorders) | 7 (7) | 7 (7)
SEXUAL/REPRODUCTIVE FUNCTION: Other (Reproductive system and breast disorders) | 2 (2) | 6 (6)
"Cardiac device implantation (pacemaker, defibrillator, etc.)" (Surgical and medical procedures) | 123 (133) | 109 (118)
"Cardiac procedure (stent, catheterization, EP study, ablation, etc.)" (Surgical and medical procedures) | 62 (76) | 66 (82)
Cardiac surgery (Surgical and medical procedures) | 28 (28) | 23 (25)
Non-cardiac surgery/Diagnostic surgery (Surgical and medical procedures) | 75 (102) | 57 (67)
SURGERY/INTRA-OPERATIVE INJURY: Other (Surgical and medical procedures) | 4 (4) | 8 (8)
Systemic embolism (Vascular disorders) | 3 (3) | 5 (5)
VASCULAR: Other (Vascular disorders) | 16 (17) | 13 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=1163) | Warfarin (N=1142)
All non-serious adverse events (General disorders) | 749 (4483) | 799 (4895)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No